CLINICAL TRIAL: NCT02356419
Title: rESP Medication With a Single Intravenous Administration and Dose Escalation to Explore the Tolerability ,Safety and Pharmacokinetic Characteristics for Healthy Subjects in the Phase Ⅰ Clinical Study
Brief Title: rESP Medication With a Single Intravenous Administration and Dose Escalation to Explore the Tolerability ,Safety and Pharmacokinetic Characteristics
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSS06
Record Dates: First submitted 2015-01-18; First posted 2015-02-05 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- experimental 0.5 ug/kg (Experimental): there are four groups in this study and healthy subjects of all groups receiving different doses of recombinant erythropoiesis stimulating protein
  Interventions: Drug: Recombinant erythropoietin stimulating protein
- experimental 1.0ug/kg (Experimental): there are four groups in this study and healthy subjects of all groups receiving different doses of recombinant erythropoiesis stimulating protein
  Interventions: Drug: Recombinant erythropoietin stimulating protein
- experimental 2.0ug/kg (Experimental): there are four groups in this study and healthy subjects of all groups receiving different doses of recombinant erythropoiesis stimulating protein
  Interventions: Drug: Recombinant erythropoietin stimulating protein
- experimental 3.0ug/kg (Experimental): there are four groups in this study and healthy subjects of all groups receiving different doses of recombinant erythropoiesis stimulating protein
  Interventions: Drug: Recombinant erythropoietin stimulating protein

INTERVENTIONS:
Drug: Recombinant erythropoietin stimulating protein — Recombinant erythropoietin stimulating protein is a high glucose medium and long-acting recombinant protein products, containing 165 amino acids by adding 3 glycosylation sites
  Other Names: Recombinant erythropoietin stimulating protein injection

SUMMARY:
The study is a single center and open test, and the dose of successive incremental method was taken. In order to determine the tolerance and safety after a single intravenous injection of different doses of rESP in healthy subjects, the investigators had this trial. On the other hand, this study is to preliminarily explore the pharmacokinetics in healthy subjects.

DETAILED DESCRIPTION:
The study is a single center and open test, and the dose of successive incremental method was taken. The study included 4 groups that is 0.5 ug/kg, 1.0ug/kg, 2.0ug/kg and 3.0ug/kg,the pharmacokinetic data (the screening period, before administration, after administration of 15, 30, 60 minutes, fourth, 8, 12, 24, 36, 48, 72 hours, seventh, 10, 14, 21, 28 days, 10 cases in each group) were collected. In order to determine the tolerance and safety after a single intravenous injection of different doses of rESP in healthy subjects, the investigators had this trial. On the other hand, this study is to preliminarily explore the pharmacokinetics in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-40 years old, male or female
2. Subjects are previously healthy, and whose physical examinations are normal 14 days ago before the screening examination
3. The BMI is 19-25Kg/m2 (BMI = weight / height2)
4. Without anemia, white blood cell and platelet counts are normal
5. Heart, lung, liver and kidney function are normal
6. Without smoke and wine hobby
7. Subjects voluntarily signing written informed consent.

Exclusion Criteria:

1. Allergic constitution or previous history of allergy of biological products;
2. Pregnant and lactating women;
3. Female subjects only take oral contraceptive pills and plan pregnancy during the clinical trials or within 3 months after administration; male subjects whose female partners plan pregnancy during the clinical trials or within 3 months after administration;
4. Female subjects received postmenopausal estrogen therapy;
5. With malignant hypertension or hypertension is poorly controlled or with previous history of thromboembolic diseases and diseases of hematopoietic system
6. Abnormal liver function ( AST or ALT is 2 times greater than the upper limit of the normal)
7. Hemoglobin is greater than or equal to 160g/L (male), 150 g/L (female)
8. The percentage of reticulocytes is greater than or equal to 3%
9. Serum iron protein <20ng/ml
10. Subjects who donated blood 90 days before being enrolled or received a blood transfusion therapy or participate in other drug test
11. subjects who received recombinant erythropoiesis stimulating protein or rHuEPO 3 months before being enrolled;
12. recombinant erythropoiesis stimulating protein antibody (RESP) or endogenous erythropoietin (EPO) antibody positive;
13. drugs known to have damage to some organs were given 3 months before being enrolled;
14. subjects whose HBsAg, HBeAg, anti-HIV, anti-HCV and syphilis antibody are positive;
15. researchers believe that other factors are not suitable for the trial

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Reticulocyte counts | 6 months
  observe the reticulocyte counts and judge whether rESP could improve anemia

SECONDARY OUTCOMES:
Hemoglobin counts | 6 months
  observe the hemoglobin counts and judge whether rESP could improve anemia

CONTACTS AND LOCATIONS:
Overall Officials: Limei Zhao, doctor, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital affiliated to China Medical University, Shenyang, Liaoning, China